CLINICAL TRIAL: NCT05795777
Title: The Frequency of Pressure Ulcers In 3rd Level Intensive Care Unıts And Determinatıon of Affectıng Risk Factors
Brief Title: Examination of the Pressure Ulcers in Intensive Care Patients.
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Refiye Akpolat, Assistant Proffesor, Kocaeli University
Other Study IDs: 0000-0001-8907-0651
Record Dates: First submitted 2023-03-09; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Pressure Ulcer; İntensive Care; Nurse's Role
Keywords: Intensive Care Unit; Pressure Ulcer; Risk Factors; Prevalence
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A pressure sore was localized skin and/or subcutaneous tissue injury, usually caused by pressure alone or a combination of shear and pressure, at bony prominences. Pressure sores, which are an indicator of the quality of health care, increase mortality, morbidity and cost. Pressure ulcers are the most common problem in intensive care patients and should be prevented. In the literature, the incidence of pressure ulcers in intensive care patients is between 1-59.9%.

A pressure sore is a localized injury to the skin and/or underlying soft tissue, usually over a bony prominence or associated with medical or other devices. This injury occurs when intense and/or prolonged pressure or pressure is accompanied by shear. Soft tissue tolerance to pressure and shear; temperature and humidity can affect nutrition, perfusion, concomitant conditions, and condition of soft tissue.

This study was carried out to determine the prevalence of pressure ulcers and influencing factors in patients hospitalized in the 3rd level intensive care unit of a university hospital.

Design: It is a descriptive, prospective, observational type study. Materials and Methods: The sample of the study consisted of 176 patients aged 18 years and above, 24 hours after hospitalization in the intensive care units of a University Hospital. Patient Information Form and Braden Scale for Predicting Pressure Ulcer Risk, Glasgow Coma Scale were used to collecting data. Statistical Package in statistical analysis for the social sciences 20.0 program was used.

DETAILED DESCRIPTION:
Due to the renovation initiated in the intensive care units, the work was started in November 2019, but the working time was extended due to the Covid 19 pandemic that developed immediately after. The sample of the study consisted of patients who met the inclusion criteria and accepted participation, among the patients who were hospitalized on Wednesday, which was determined as the middle of each week, between November 2019 and February 2021 in the 3rd-level intensive care units of a university hospital.

Data Collection: "Personal Information Form" prepared by the researcher as a result of the literature review for data collection, "Braden Scale for Predicting Pressure Ulcer Risk" for evaluating pressure ulcers, "Glasgow Coma Score" for evaluating patient's consciousness status, and ulcer used by National Pressure Ulcer Advisory Panel and European Pressure Ulcer Advisory Panel staging classification was used.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* Hospitalized in the 3rd step intensive care unit
* Being hospitalized for at least 24 hours
* No pressure ulcers on the first hospitalization

Exclusion Criteria:

* hospitalization time not exceeding 24 hours

Ages: 18 Years to 92 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in 3rd level intensive care units
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Data collection from patients | 15 minutes
  The sample of the study consisted of patients who were hospitalized in the tertiary intensive care unit of a university hospital between November 2019 and February 2021, who met the inclusion criteria and accepted to participate in the study. Data were collected from patients every Wednesday, which was determined as the middle of the week. Patients were evaluated with the Braden Scale for Predicting Pressure Ulcer Risk. The total score of the scale varies between 6-23 points. As the scores obtained from the scale decrease, the risk of developing pressure ulcers increases. A scale score of 9 or less indicates a high risk, and a scale score of 19-23 indicates no risk.
  Data collection from each patient took 15 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Refiye Akpolat, Principal Investigator — Kocaeli Healt and Tecnology University
Locations (1):
- Kocaeli Healt and Tecnology University, Kocaeli, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No